CLINICAL TRIAL: NCT04386616
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of MSTT1041A or UTTR1147A in Patients With Severe COVID-19 Pneumonia
Brief Title: A Study to Evaluate the Safety and Efficacy of MSTT1041A (Astegolimab) or UTTR1147A in Patients With Severe COVID-19 Pneumonia
Acronym: COVASTIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA42469; 2020-002713-17 (EudraCT Number); OT number: HHSO100201800036C (Other Grant/Funding Number: Biomedical Advanced Research and Development Authority)
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — astegolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- All Placebo (Placebo Comparator): Participants randomized to this arm received one intravenous (IV) infusion of either MSTT1041A-matched placebo or UTTR1147A-matched placebo on Day 1. A second IV infusion of either MSTT1041A-matched placebo or UTTR1147A-matched placebo (same placebo as the first infusion) was given on Day 15 if the participant remained hospitalized with a requirement for supplemental oxygen. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
  Interventions: Drug: MSTT1041A-matched Placebo; Drug: UTTR1147A-matched Placebo
- MSTT1041A (Experimental): Participants randomized to this arm received one intravenous (IV) infusion of MSTT1041A 700 milligrams (mg) on Day 1. A second IV dose of MSTT1041A 350 mg was given on Day 15 if the participant remained hospitalized with a requirement for supplemental oxygen. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
  Interventions: Drug: MSTT1041A
- UTTR1147A (Experimental): Participants randomized to this arm received one intravenous (IV) infusion of UTTR1147A 90 micrograms/kilogram body weight (μg/kg) on Day 1. A second IV dose of UTTR1147A 90 μg/kg was given on Day 15 if the participant remained hospitalized with a requirement for supplemental oxygen. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
  Interventions: Drug: UTTR1147A

INTERVENTIONS:
Drug: MSTT1041A — Participants received one intravenous (IV) infusion of MSTT1041A 700 milligrams (mg) on Day 1. A second IV dose of MSTT1041A 350 mg was given on Day 15 if the participant remained hospitalized with a requirement for supplemental oxygen.
  Other Names: Astegolimab; RG6149; RO7187807
  Arms: MSTT1041A
Drug: MSTT1041A-matched Placebo — Participants received up to 2 intravenous infusions of MSTT1041A-matched placebo.
  Arms: All Placebo
Drug: UTTR1147A — Participants received one intravenous (IV) infusion of UTTR1147A 90 micrograms/kilogram body weight (μg/kg) on Day 1. A second IV dose of UTTR1147A 90 μg/kg was given on Day 15 if the participant remained hospitalized with a requirement for supplemental oxygen.
  Other Names: Efmarodocokin alfa; RG7880; RO7021610; IL-22Fc
  Arms: UTTR1147A
Drug: UTTR1147A-matched Placebo — Participants received up to 2 intravenous infusions of UTTR1147A-matched placebo.
  Arms: All Placebo

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of MSTT1041A (astegolimab) compared with placebo and of UTTR1147A compared with placebo, in combination with standard of care (SOC), in patients hospitalized with severe coronavirus disease 2019 (COVID-19) pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with COVID-19 pneumonia confirmed per WHO criteria (including a positive PCR of any specimen; e.g., respiratory, blood, urine, stool, other bodily fluid) and evidenced by chest X-ray or CT scan
* Peripheral capillary oxygen saturation (SpO2) ≤93% (on room air or supplemental oxygen) or partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2) ≤300 millimetres of mercury (mmHg) or requiring supplemental oxygen to maintain SpO2 >93% or requirement for supplemental oxygen to maintain SpO2 at an acceptable level per local standard of care

Exclusion Criteria:

* Pregnant or breastfeeding, or positive pregnancy test at screening
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Participating in another clinical drug trial
* Treatment with investigational therapy (other than for COVID-19) within 5 half-lives or 30 days (whichever is longer) prior to initiation of study drug
* Use of Janus kinase (JAK) inhibitor within 30 days or 5 drug elimination half-lives (whichever is longer) prior to screening
* Have received high-dose systemic corticosteroids (≥1 mg/kg/day methylprednisolone or equivalent) within 72 hours prior to Day 1
* Known HIV infection with CD4 <200 cells/microlitre (uL) or <14% of all lymphocytes
* ALT or AST >10 times the upper limit of normal (ULN) detected at screening
* History of anaplastic large-cell lymphoma or mantle-cell lymphoma
* History of cancer within the previous 5 years unless it has been adequately treated and considered cured or remission-free in the investigator's judgment
* Clinical evidence of active or unstable cardiovascular disease (e.g., acute myocardial ischemia or decompensated heart failure), as determined by investigator assessment, ECG, laboratory assessment, or echocardiographic data
* History of moderate or severe allergic, anaphylactic, or anaphylactoid reactions or hypersensitivity to any component of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (41):
- United States (24):
  - University of Arkansas For Medical Sciences, Little Rock, Arkansas
  - eStudySite - Chula Vista - PPDS, Chula Vista, California
  - eStudySite, La Mesa, California
  - Torrance Memorial Medical Center, Torrance, California
  - Denver Health Medical Center, Denver, Colorado
  - Bay Pines VA Medical Center - NAVREF, Bay Pines, Florida
  - WellStar Research Institute, Marietta, Georgia
  - DM Clinical Research - Alexandria Cardiology Clinic - ERN - PPDS, Alexandria, Louisiana
  - MedPharmics, Metairie, Louisiana
  - Southeast Louisiana Veterans Health Care System - NAVREF, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - St. Joseph'S Regional Medical Center, Paterson, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Albany Medical Center, Albany, New York
  - Staten Island University Hospital; Department of Pharmacy, Staten Island, New York
  - Lincoln Medical Mental Health Center, The Bronx, New York
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Providence Portland Medical Center; Investigational Drug Services/Regional Research, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Parkland Health & Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - MultiCare Institute for Research and Innovation; Clinic/Outpatient Facility, Tacoma, Washington
- Brazil (6):
  - Instituto de Pesquisa Clinica Evandro Chagas FIOCRUZ, Rio de Janeiro, Rio de Janeiro
  - Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital E Maternidade Celso Pierro PUCCAMP, Campinas, São Paulo
  - Hospital de Base Da Faculdade de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Instituto do Coração - HCFMUSP, São Paulo, São Paulo
- Mexico (5):
  - Nuevo Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, México
  - Instituto Nacional De Enfermedades Respiratorias INER National Institute of Respiratory Diseases, México
  - Hospital General de Tijuana, Tijuana
- Spain (6):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Costa del Sol; Servicio de Oncologia, Marbella, Malaga
  - Hospital del Mar, Barcelona
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Clinico Universitario Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Waters M, McKinnell JA, Kalil AC, Martin GS, Buchman TG, Theess W, Yang X, Lekkerkerker AN, Staton T, Rosenberger CM, Pappu R, Wang Y, Zhang W, Brooks L, Cheung D, Galanter J, Chen H, Mohan D, Peck MC; COVID-astegolimab-interleukin (IL) (COVASTIL) Study Group. Astegolimab or Efmarodocokin Alfa in Patients With Severe COVID-19 Pneumonia: A Randomized, Phase 2 Trial. Crit Care Med. 2023 Jan 1;51(1):103-116. doi: 10.1097/CCM.0000000000005716. Epub 2022 Nov 14. PMID 36519984

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Started | 134 | 130 | 132
Received at Least One Dose of Study Drug (Safety Population) | 134 (In this arm, 68 and 66 participants received MSTT1041A-matched placebo and UTTR1147A-matched placebo, respectively.) | 130 | 132
Completed Both Doses of Study Drug at Day 15 | 31 | 27 | 25
Completed | 104 | 95 | 104
Not Completed | 30 | 35 | 28
Not completed — Death | 22 | 22 | 21
Not completed — Lost to Follow-up | 5 | 8 | 6
Not completed — Withdrawal by Subject | 2 | 4 | 1
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) Population: all participants randomized in the study who received at least one dose of study drug, with participants grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | All Placebo | MSTT1041A | UTTR1147A | Total
Number analyzed (Participants) | 134 | 130 | 132 | 396
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (13.5) | 57.3 (13.4) | 57.8 (12.6) | 57.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 56 | 52 | 153
  Male | 89 | 74 | 80 | 243
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 72 | 70 | 219
  Not Hispanic or Latino | 53 | 53 | 58 | 164
  Unknown or Not Reported | 4 | 5 | 4 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 0 | 6
  Asian | 6 | 4 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 4 | 1 | 5
  Black or African American | 10 | 7 | 10 | 27
  White | 92 | 87 | 89 | 268
  Unknown | 24 | 24 | 27 | 75
Region of Enrollment [Count of Participants; unit: Participants] — Regional enrollment included the following countries: North America = Mexico and United States; South America = Brazil; and Western Europe = Spain. This was one of the two stratification factors at randomization.
  Participants
    North America | 99 | 97 | 97 | 293
    South America | 19 | 20 | 20 | 59
    Western Europe | 16 | 13 | 15 | 44
Country of Enrollment [Count of Participants; unit: Participants]
  Brazil | 19 | 20 | 20 | 59
  Mexico | 14 | 23 | 17 | 54
  Spain | 16 | 13 | 15 | 44
  United States | 85 | 74 | 80 | 239
Mechanical Ventilation Required (Yes/No) [Count of Participants; unit: Participants] — This was one of the two stratification factors at randomization.
  Participants
    Yes, Baseline Mechanical Ventilation | 12 | 13 | 11 | 36
    No Baseline Mechanical Ventilation | 122 | 117 | 121 | 360
Clinical Status Score at Baseline [Count of Participants; unit: Participants] — The 7 categories of the clinical status ordinal scale are defined as follows: 1. Discharged (or "ready for discharge"); 2. Non-Intensive Care Unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen; 3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen; 4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen; 5. ICU, requiring intubation and mechanical ventilation; 6. ICU, requiring ECMO or mechanical ventilation and additional organ support; 7. Death
  Participants
    Clinical Status Score of 1 | 0 | 0 | 0 | 0
    Clinical Status Score of 2 | 3 | 4 | 1 | 8
    Clinical Status Score of 3 | 47 | 49 | 57 | 153
    Clinical Status Score of 4 | 71 | 64 | 63 | 198
    Clinical Status Score of 5 | 10 | 8 | 8 | 26
    Clinical Status Score of 6 | 3 | 4 | 2 | 9
    Clinical Status Score of 7 | 0 | 0 | 0 | 0
    Clinical Status Score Not Available | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery, Defined as the Time to a Clinical Status Score of 1 or 2 on the 7-Category Ordinal Scale (Whichever Occurs First) by Day 28
Description: The time to recovery was defined as the time from baseline to a clinical status score of 1 or 2 on the 7-category ordinal scale (whichever occurs first); clinical status scores are defined as follows: 1. Discharged (or "ready for discharge" as evidenced by normal body temperature and respiratory rate, and stable oxygen saturation on ambient air or ≤2 Litres supplemental oxygen); 2. Non-Intensive Care Unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen; 3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen; 4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen; 5. ICU, requiring intubation and mechanical ventilation; 6. ICU, requiring extracorporeal membrane oxygenation (ECMO) or mechanical ventilation and additional organ support (e.g., vasopressors, renal replacement therapy); 7. Death.
Time Frame: From Baseline up to 28 days
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Days | 10.0 [8.0 to 14.0] | 11.0 [9.0 to 14.0] | 10.0 [8.0 to 13.0]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.9266, Unstratified Log Rank — p<0.05 threshold for statistical significance; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.75 to 1.36] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.3570, Unstratified Log Rank — p<0.05 threshold for statistical significance; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.86 to 1.54] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.9812, Stratified Log Rank — p<0.05 threshold for statistical significance; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.74 to 1.36] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.5151, Stratified Log Rank — p<0.05 threshold for statistical significance; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.82 to 1.49] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

2. Secondary Outcome: Time to Improvement of at Least 2 Categories Relative to Baseline on a 7-Category Ordinal Scale of Clinical Status by Day 28
Description: The 7 categories of the clinical status ordinal scale are defined as follows: 1. Discharged (or "ready for discharge" as evidenced by normal body temperature and respiratory rate, and stable oxygen saturation on ambient air or ≤2 Litres supplemental oxygen); 2. Non-Intensive Care Unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen; 3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen; 4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen; 5. ICU, requiring intubation and mechanical ventilation; 6. ICU, requiring ECMO or mechanical ventilation and additional organ support (e.g., vasopressors, renal replacement therapy); 7. Death
Time Frame: From Baseline up to 28 days
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Days | 10.0 [8.0 to 14.0] | 11.0 [9.0 to 13.0] | 10.0 [8.0 to 12.0]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.8373, Unstratified Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.77 to 1.39] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.3396, Unstratified Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.86 to 1.55] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.8619, Stratified Log Rank; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.76 to 1.39] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.4913, Stratified Log Rank; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.82 to 1.50] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

3. Secondary Outcome: Time to Hospital Discharge or "Ready for Discharge" by Day 28
Description: Hospital discharge is category number 1 out of the 7 categories of the clinical status ordinal scale, and it is defined as follows: 1. Discharged (or "ready for discharge" as evidenced by normal body temperature and respiratory rate, and stable oxygen saturation on ambient air or ≤2 Litres supplemental oxygen).
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Days | 10.0 [8.0 to 14.0] | 11.0 [9.0 to 13.0] | 10.0 [8.0 to 13.0]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.4711, Unstratified Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.83 to 1.49] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.3135, Unstratified Log Rank; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.87 to 1.56] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.5735, Stratified Log Rank; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.81 to 1.48] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.5973, Stratified Log Rank; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.80 to 1.46] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

4. Secondary Outcome: Duration of Supplemental Oxygen by Day 28
Description: Duration of supplemental oxygen was defined as the number of days during the 28-day treatment period when the participant is alive and receives "Supplemental Oxygen or other forms of ventilation", as recorded in the Vital Signs and Oxygen Saturation form. For each participant, the duration of multiple non-consecutive periods during which the participant received supplemental oxygen was summed. For any days prior to Day 28 where status of supplemental oxygen use was missing, the last known status was to be carried forward.
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Days | 18.00 [13.00 to 27.00] | 17.00 [11.00 to 27.00] | 13.50 [10.00 to 21.00]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.5304, Van Elteren; Median Difference (Net) = -1.00 — The median difference was calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.5058, Van Elteren; Median Difference (Net) = -4.50 — The median difference was calculated as the UTT1147A Arm minus the Placebo Arm

5. Secondary Outcome: Percentage of Participants Alive and Free of Respiratory Failure by Day 28
Description: Respiratory failure was defined as requiring non-invasive ventilation, high-flow oxygen, mechanical ventilation, or extracorporeal membrane oxygenation [ECMO]).
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Percentage of participants | 38.1 [29.47 to 46.65] | 39.2 [30.45 to 48.01] | 40.2 [31.41 to 48.89]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.8451, Chi-squared; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.64 to 1.72] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.7267, Chi-squared; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.67 to 1.79] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.8458, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.63 to 1.79] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.7907, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.64 to 1.81] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

6. Secondary Outcome: Clinical Status Score at Day 14, Assessed Using a 7-Category Ordinal Scale
Description: The clinical status scores of the 7 category ordinal scale are defined as follows: 1. Discharged (or "ready for discharge" as evidenced by normal body temperature and respiratory rate, and stable oxygen saturation on ambient air or ≤2 Litres supplemental oxygen); 2. Non-Intensive Care Unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen; 3. Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen; 4. ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen; 5. ICU, requiring intubation and mechanical ventilation; 6. ICU, requiring ECMO or mechanical ventilation and additional organ support (e.g., vasopressors, renal replacement therapy); 7. Death
Time Frame: Day 14
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Score on a scale | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 4.0]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.5273, Van Elteren; Median Difference (Final Values) = 0.0 — The median difference was calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.6515, Van Elteren; Median Difference (Final Values) = 0.0 — The median difference was calculated as the UTT1147A Arm minus the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.5475, Proportional Odds Model; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.71 to 1.91] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.5652, Proportional Odds Model; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.71 to 1.89] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

7. Secondary Outcome: Clinical Status Score at Day 28, Assessed Using a 7-Category Ordinal Scale
Description: as for outcome 6
Time Frame: Day 28
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Score on a scale | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.3401, Van Elteren; Median Difference (Final Values) = 0.0 — The median difference was calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.4676, Van Elteren; Median Difference (Final Values) = 0.0 — The median difference was calculated as the UTT1147A Arm minus the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.3408, Proportional Odds Model; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.75 to 2.29] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.3320, Proportional Odds Model; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.76 to 2.29] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

8. Secondary Outcome: Percentage of Participants Needing Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO) by Day 28
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Percentage of participants | 24.6 [16.96 to 32.29] | 28.5 [20.32 to 36.60] | 24.2 [16.55 to 31.93]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; Difference in percentage of participants = 3.83, 95% CI 2-sided [-7.57 to 15.24] — The difference in percentage of participants was calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; Difference in percentage of participants = -0.38, 95% CI 2-sided [-11.46 to 10.70] — The difference in percentage of participants was calculated as the UTTR1147A Arm minus the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.4804, Chi-squared; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.70 to 2.10] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.9418, Chi-squared; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.56 to 1.71] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 5: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.4988, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.68 to 2.44] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 6: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.9043, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.54 to 1.96] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

9. Secondary Outcome: Number of Ventilator-Free Days by Day 28
Description: The number of ventilator-free days was defined as the number of days during the 28-day treatment period when the participant is alive and without need for invasive mechanical ventilation. For any day during Day 1 and Day 28, if invasive mechanical ventilation or ECMO was recorded for any part of the day ( >= 12 hours during mechanical invasive ventilation for patients with tracheostomy), the day was not to be counted as a ventilator-free day; otherwise, the day was to be counted. For any days prior to Day 28 where status of mechanical ventilator was missing, the last known status was to be carried forward. The total number of days was the sum of all ventilator-free days, regardless of whether the days occurred consecutively or in nonconsecutive intervals.
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Days | 28.0 [20.00 to 28.00] | 28.0 [20.00 to 28.00] | 28.0 [23.50 to 28.00]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.8007, Van Elteren; Median Difference (Net) = 0.0 — Median difference was calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.8633, Van Elteren; Median Difference (Net) = 0.0 — Median difference was calculated as the UTTR1147A Arm minus the Placebo Arm

10. Secondary Outcome: Percentage of Participants With an Intensive Care Unit (ICU) Stay by Day 28
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Percentage of participants | 58.2 [49.48 to 66.93] | 54.6 [45.67 to 63.56] | 46.2 [37.33 to 55.10]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; Difference in percentage of participants = -3.59, 95% CI 2-sided [-16.31 to 9.12] — The difference in percentage of participants was calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; Difference in percentage of participants = -12.00, 95% CI 2-sided [-24.67 to 0.67] — The difference in percentage of participants was calculated as the UTTR1147A Arm minus the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.5560, Chi-squared; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.53 to 1.41] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.0502, Chi-squared; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.38 to 1.00] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 5: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.7002, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.51 to 1.60] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 6: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.0448, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.32 to 0.99] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

11. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay by Day 28
Description: Duration of ICU stay was calculated as the total number of hours (expressed in days) spent in ICU up to and inclusive of 28 days. ICU duration was derived from the ICU Stay Information Log using the difference between ICU discharge date/time and ICU admission date/time. If ICU admission occurred before randomization, the ICU duration was to be counted from the date of dosing. Partial admission and discharge date/time were to be imputed following a conservative approach. For each participant, durations of multiple ICU stays were to be summed.
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Days | 3.10 [0.00 to 5.23] | 2.62 [0.00 to 6.02] | 0.00 [0.00 to 2.14]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.4845, Van Elteren; Median Difference (Net) = -0.48 — Median difference was calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.0570, Van Elteren; Median Difference (Net) = -3.10 — Median difference was calculated as the UTTR1147A Arm minus the Placebo Arm

12. Secondary Outcome: Time to Clinical Failure by Day 28, Defined as the Time to Death, Mechanical Ventilation, ICU Admission, or Withdrawal of Care (Whichever Occurs First)
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Days | NA [13.0 to NA] — The median and upper limit of the interquartile range could not be estimated because an insufficient number of clinical failure events had occurred. | NA [9.0 to NA] — The median and upper limit of the interquartile range could not be estimated because an insufficient number of clinical failure events had occurred. | NA [NA to NA] — The median and lower and upper limits of the interquartile range could not be estimated because an insufficient number of clinical failure events had occurred.
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.4456, Unstratified Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.76 to 1.88] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.7213, Unstratified Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.57 to 1.48] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.3963, Stratified Log Rank; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.77 to 1.96] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.9174, Stratified Log Rank; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.60 to 1.58] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

13. Secondary Outcome: Percentage of Participants Who Died by Day 14
Time Frame: Up to Day 14
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Percentage of participants | 6.0 [1.59 to 10.35] | 8.5 [3.29 to 13.63] | 8.3 [3.24 to 13.43]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Other; Difference in Mortality Rates = 2.49, 95% CI 2-sided [-4.51 to 9.49] — The difference in mortality rates is calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Other; Difference in Mortality Rates = 2.36, 95% CI 2-sided [-4.58 to 9.31] — The difference in mortality rates is calculated as the UTTR1147A Arm minus the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.4336, Chi-squared; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.57 to 3.74] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.4543, Chi-squared; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.56 to 3.68] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 5: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.4900, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.54 to 3.97] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 6: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.3595, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.58 to 4.28] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

14. Secondary Outcome: Percentage of Participants Who Died by Day 28
Time Frame: Up to Day 28
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Percentage of participants | 11.2 [5.48 to 16.91] | 14.6 [8.16 to 21.07] | 12.9 [6.79 to 18.97]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Other; Difference in Mortality Rates = 3.42, 95% CI 2-sided [-5.42 to 12.26] — The difference in mortality rates is calculated as the MSTT1041A Arm minus the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Other; Difference in Mortality Rates = 1.68, 95% CI 2-sided [-6.89 to 10.26] — The difference in mortality rates is calculated as the UTTR1147A Arm minus the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.4067, Chi-squared; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.66 to 2.80] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.6728, Chi-squared; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.56 to 2.46] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 5: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.5495, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.62 to 2.87] — The odds ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 6: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.5551, Cochran-Mantel-Haenszel; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.57 to 2.71] — The odds ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

15. Secondary Outcome: Time to Clinical Improvement, Defined as a National Early Warning Score 2 (NEWS2) Aggregate Score of ≤2 Maintained for 24 Hours
Description: The National Early Warning Score 2 (NEWS2) is a system for scoring the physiological measurements that are routinely recorded at the patient's bedside. Its purpose is to identify acutely ill patients. The NEWS2 scoring system measures 7 physiological parameters: respiration rate, peripheral capillary oxygen saturation, breathing air or supplementary oxygen, systolic blood pressure, pulse rate, level of consciousness or new-onset confusion, and body temperature. A score of 0, 1, 2, or 3 is allocated to each parameter (except for air or oxygen, with respective scores of 0 and 2); a higher score means the parameter is further from the normal range. The scores for each parameter are then summed (with an aggregate score ranging from 0 to 20), and a higher aggregate score indicates a worse clinical condition of the patient, thus indicating the need for a more urgent clinical response.
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Days | 5.5 [4.0 to 7.0] | 6.0 [4.0 to 8.0] | 6.0 [3.0 to 9.0]
Statistical Analysis 1: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.3831, Unstratified Log Rank; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.71 to 2.40] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 2: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.5925, Unstratified Log Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.65 to 2.15] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm
Statistical Analysis 3: Comparison: All Placebo vs MSTT1041A; Test type: Superiority; p = 0.7487, Stratified Log Rank; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.60 to 2.05] — The hazard ratio was calculated as the MSTT1041A Arm relative to the Placebo Arm
Statistical Analysis 4: Comparison: All Placebo vs UTTR1147A; Test type: Superiority; p = 0.6092, Stratified Log Rank; The analysis was adjusted for the baseline characteristics of region of enrollment and need for mechanical ventilation; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.63 to 2.21] — The hazard ratio was calculated as the UTTR1147A Arm relative to the Placebo Arm

16. Secondary Outcome: Safety Summary of the Number of Participants With at Least One Adverse Event, With Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Description: The terms "severe" and "serious" are not synonymous with respect to an adverse event (AE). Severity refers to the intensity of an AE (rated according to NCI-CTCAE v5.0 criteria or, if not listed, the following scale: Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to AE), whereas a serious AE (SAE) is a significant medical event (per standard SAE criteria), such as a life-threatening or fatal AE or an AE that prolongs inpatient hospitalization. Severity and seriousness were independently assessed by the investigator for each AE that was recorded. The investigator also assessed each AE for whether the event was considered to be related to the study drug.
Time Frame: From Baseline until study completion/discontinuation (up to 60 days)
Population: Safety Population: participants who received at least one dose of study drug, with participants grouped according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Participants
  Any Adverse Event (AE) | 87 | 85 | 95
  AE with Fatal Outcome | 23 | 23 | 21
  Serious AE (SAE) | 38 | 38 | 34
  SAE Leading to Withdrawal from Treatment | 2 | 2 | 1
  SAE Leading to Dose Modification/Interruption | 0 | 0 | 0
  Related SAE | 0 | 2 | 3
  AE Leading to Withdrawal from Treatment | 4 | 3 | 3
  AE Leading to Dose Modification/Interruption | 0 | 0 | 0
  Related AE | 15 | 12 | 25
  Related AE Leading to Withdrawal from Treatment | 0 | 0 | 1
  Related AE Leading to Dose Modification/Interruption | 0 | 0 | 0
  Grade 3-5 AE | 43 | 46 | 41

17. Secondary Outcome: Number of Participants With Clinical Laboratory Test Abnormalities by Highest NCI-CTCAE Grade Post-Baseline
Description: Clinical laboratory tests were performed over the course of the study and the grading of any abnormal values outside of the normal range (High or Low) was based on the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0); the higher the grade, the greater the lab parameter deviated from the normal range. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. SGPT/ALT = alanine aminotransferase; SGOT/AST = aspartate aminotransferase; INR = international normalized ratio; aPTT = activated partial thromboplastin time
Time Frame: From Baseline up to 60 days
Population: Safety Population: participants who received at least one dose of study drug, with participants grouped according to the treatment received. Only participants with both a baseline assessment and at least one post-baseline assessment per parameter were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Participants
  Albumin, Low - Any Grade: number analyzed (Participants) | 133 | 129 | 131
  Albumin, Low - Any Grade | 103 | 105 | 118
  Albumin, Low - Grade 1: number analyzed (Participants) | 133 | 129 | 131
  Albumin, Low - Grade 1 | 32 | 36 | 40
  Albumin, Low - Grade 2: number analyzed (Participants) | 133 | 129 | 131
  Albumin, Low - Grade 2 | 56 | 58 | 66
  Albumin, Low - Grade 3: number analyzed (Participants) | 133 | 129 | 131
  Albumin, Low - Grade 3 | 15 | 11 | 12
  Alkaline Phosphatase, High - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Alkaline Phosphatase, High - Any Grade | 20 | 23 | 24
  Alkaline Phosphatase, High - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Alkaline Phosphatase, High - Grade 1 | 14 | 22 | 22
  Alkaline Phosphatase, High - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Alkaline Phosphatase, High - Grade 2 | 5 | 1 | 1
  Alkaline Phosphatase, High - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Alkaline Phosphatase, High - Grade 3 | 1 | 0 | 1
  SGPT/ALT, High - Any Grade: number analyzed (Participants) | 132 | 129 | 132
  SGPT/ALT, High - Any Grade | 60 | 48 | 60
  SGPT/ALT, High - Grade 1: number analyzed (Participants) | 132 | 129 | 132
  SGPT/ALT, High - Grade 1 | 48 | 37 | 47
  SGPT/ALT, High - Grade 2: number analyzed (Participants) | 132 | 129 | 132
  SGPT/ALT, High - Grade 2 | 5 | 7 | 7
  SGPT/ALT, High - Grade 3: number analyzed (Participants) | 132 | 129 | 132
  SGPT/ALT, High - Grade 3 | 5 | 3 | 5
  SGPT/ALT, High - Grade 4: number analyzed (Participants) | 132 | 129 | 132
  SGPT/ALT, High - Grade 4 | 2 | 1 | 1
  SGOT/AST, High - Any Grade: number analyzed (Participants) | 133 | 129 | 131
  SGOT/AST, High - Any Grade | 47 | 38 | 44
  SGOT/AST, High - Grade 1: number analyzed (Participants) | 133 | 129 | 131
  SGOT/AST, High - Grade 1 | 40 | 30 | 36
  SGOT/AST, High - Grade 2: number analyzed (Participants) | 133 | 129 | 131
  SGOT/AST, High - Grade 2 | 4 | 5 | 4
  SGOT/AST, High - Grade 3: number analyzed (Participants) | 133 | 129 | 131
  SGOT/AST, High - Grade 3 | 0 | 2 | 2
  SGOT/AST, High - Grade 4: number analyzed (Participants) | 133 | 129 | 131
  SGOT/AST, High - Grade 4 | 3 | 1 | 2
  Calcium, Low - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Calcium, Low - Any Grade | 73 | 82 | 84
  Calcium, Low - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Calcium, Low - Grade 1 | 34 | 47 | 48
  Calcium, Low - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Calcium, Low - Grade 2 | 31 | 26 | 29
  Calcium, Low - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Calcium, Low - Grade 3 | 5 | 7 | 4
  Calcium, Low - Grade 4: number analyzed (Participants) | 133 | 130 | 132
  Calcium, Low - Grade 4 | 3 | 2 | 3
  Calcium, High - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Calcium, High - Any Grade | 5 | 2 | 4
  Calcium, High - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Calcium, High - Grade 1 | 5 | 2 | 4
  Creatinine, High - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Creatinine, High - Any Grade | 24 | 39 | 29
  Creatinine, High - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Creatinine, High - Grade 1 | 6 | 11 | 8
  Creatinine, High - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Creatinine, High - Grade 2 | 11 | 24 | 15
  Creatinine, High - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Creatinine, High - Grade 3 | 7 | 3 | 5
  Creatinine, High - Grade 4: number analyzed (Participants) | 133 | 130 | 132
  Creatinine, High - Grade 4 | 0 | 1 | 1
  Fibrinogen, Low - Any Grade: number analyzed (Participants) | 125 | 122 | 130
  Fibrinogen, Low - Any Grade | 7 | 3 | 1
  Fibrinogen, Low - Grade 1: number analyzed (Participants) | 125 | 122 | 130
  Fibrinogen, Low - Grade 1 | 1 | 1 | 0
  Fibrinogen, Low - Grade 2: number analyzed (Participants) | 125 | 122 | 130
  Fibrinogen, Low - Grade 2 | 3 | 2 | 0
  Fibrinogen, Low - Grade 3: number analyzed (Participants) | 125 | 122 | 130
  Fibrinogen, Low - Grade 3 | 2 | 0 | 0
  Fibrinogen, Low - Grade 4: number analyzed (Participants) | 125 | 122 | 130
  Fibrinogen, Low - Grade 4 | 1 | 0 | 1
  Glucose, Low - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Glucose, Low - Any Grade | 8 | 11 | 12
  Glucose, Low - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Glucose, Low - Grade 1 | 6 | 6 | 9
  Glucose, Low - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Glucose, Low - Grade 2 | 1 | 5 | 0
  Glucose, Low - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Glucose, Low - Grade 3 | 1 | 0 | 2
  Glucose, Low - Grade 4: number analyzed (Participants) | 133 | 130 | 132
  Glucose, Low - Grade 4 | 0 | 0 | 1
  Hemoglobin, Low - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Hemoglobin, Low - Any Grade | 77 | 72 | 78
  Hemoglobin, Low - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Hemoglobin, Low - Grade 1 | 43 | 47 | 46
  Hemoglobin, Low - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Hemoglobin, Low - Grade 2 | 17 | 17 | 21
  Hemoglobin, Low - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Hemoglobin, Low - Grade 3 | 17 | 8 | 11
  Hemoglobin, High - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Hemoglobin, High - Any Grade | 9 | 7 | 5
  Hemoglobin, High - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Hemoglobin, High - Grade 1 | 9 | 6 | 5
  Hemoglobin, High - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Hemoglobin, High - Grade 3 | 0 | 1 | 0
  Lymphocytes, Absolute Count (Abs), Low - Any Grade: number analyzed (Participants) | 100 | 91 | 93
  Lymphocytes, Absolute Count (Abs), Low - Any Grade | 61 | 45 | 48
  Lymphocytes, Abs, Low - Grade 1: number analyzed (Participants) | 100 | 91 | 93
  Lymphocytes, Abs, Low - Grade 1 | 14 | 9 | 11
  Lymphocytes, Abs, Low - Grade 2: number analyzed (Participants) | 100 | 91 | 93
  Lymphocytes, Abs, Low - Grade 2 | 23 | 17 | 23
  Lymphocytes, Abs, Low - Grade 3: number analyzed (Participants) | 100 | 91 | 93
  Lymphocytes, Abs, Low - Grade 3 | 23 | 18 | 11
  Lymphocytes, Abs, Low - Grade 4: number analyzed (Participants) | 100 | 91 | 93
  Lymphocytes, Abs, Low - Grade 4 | 1 | 1 | 3
  Lymphocytes, Abs, High - Any Grade: number analyzed (Participants) | 100 | 91 | 93
  Lymphocytes, Abs, High - Any Grade | 4 | 4 | 1
  Lymphocytes, Abs, High - Grade 2: number analyzed (Participants) | 100 | 91 | 93
  Lymphocytes, Abs, High - Grade 2 | 4 | 4 | 1
  Neutrophils, Total (Abs), Low - Any Grade: number analyzed (Participants) | 100 | 91 | 93
  Neutrophils, Total (Abs), Low - Any Grade | 5 | 3 | 1
  Neutrophils, Total (Abs), Low - Grade 1: number analyzed (Participants) | 100 | 91 | 93
  Neutrophils, Total (Abs), Low - Grade 1 | 4 | 3 | 0
  Neutrophils, Total (Abs), Low - Grade 2: number analyzed (Participants) | 100 | 91 | 93
  Neutrophils, Total (Abs), Low - Grade 2 | 1 | 0 | 1
  Platelets, Low - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Platelets, Low - Any Grade | 17 | 17 | 12
  Platelets, Low - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Platelets, Low - Grade 1 | 14 | 15 | 9
  Platelets, Low - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Platelets, Low - Grade 2 | 2 | 0 | 2
  Platelets, Low - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Platelets, Low - Grade 3 | 1 | 1 | 0
  Platelets, Low - Grade 4: number analyzed (Participants) | 133 | 130 | 132
  Platelets, Low - Grade 4 | 0 | 1 | 1
  Potassium, Low - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Potassium, Low - Any Grade | 29 | 19 | 25
  Potassium, Low - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Potassium, Low - Grade 2 | 25 | 18 | 23
  Potassium, Low - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Potassium, Low - Grade 3 | 4 | 1 | 2
  Potassium, High - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Potassium, High - Any Grade | 15 | 25 | 16
  Potassium, High - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Potassium, High - Grade 1 | 7 | 19 | 12
  Potassium, High - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Potassium, High - Grade 2 | 5 | 3 | 3
  Potassium, High - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Potassium, High - Grade 3 | 2 | 3 | 1
  Potassium, High - Grade 4: number analyzed (Participants) | 133 | 130 | 132
  Potassium, High - Grade 4 | 1 | 0 | 0
  INR, High - Any Grade: number analyzed (Participants) | 126 | 125 | 130
  INR, High - Any Grade | 71 | 69 | 75
  INR, High - Grade 1: number analyzed (Participants) | 126 | 125 | 130
  INR, High - Grade 1 | 60 | 61 | 67
  INR, High - Grade 2: number analyzed (Participants) | 126 | 125 | 130
  INR, High - Grade 2 | 9 | 8 | 6
  INR, High - Grade 3: number analyzed (Participants) | 126 | 125 | 130
  INR, High - Grade 3 | 2 | 0 | 2
  aPTT, High - Any Grade: number analyzed (Participants) | 121 | 126 | 128
  aPTT, High - Any Grade | 47 | 42 | 42
  aPTT, High - Grade 1: number analyzed (Participants) | 121 | 126 | 128
  aPTT, High - Grade 1 | 38 | 35 | 36
  aPTT, High - Grade 2: number analyzed (Participants) | 121 | 126 | 128
  aPTT, High - Grade 2 | 6 | 5 | 3
  aPTT, High - Grade 3: number analyzed (Participants) | 121 | 126 | 128
  aPTT, High - Grade 3 | 3 | 2 | 3
  Sodium, Low - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Sodium, Low - Any Grade | 67 | 58 | 58
  Sodium, Low - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Sodium, Low - Grade 1 | 60 | 50 | 51
  Sodium, Low - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Sodium, Low - Grade 2 | 6 | 6 | 7
  Sodium, Low - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Sodium, Low - Grade 3 | 1 | 1 | 0
  Sodium, Low - Grade 4: number analyzed (Participants) | 133 | 130 | 132
  Sodium, Low - Grade 4 | 0 | 1 | 0
  Sodium, High - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Sodium, High - Any Grade | 17 | 16 | 23
  Sodium, High - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Sodium, High - Grade 1 | 11 | 10 | 21
  Sodium, High - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Sodium, High - Grade 2 | 5 | 5 | 1
  Sodium, High - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Sodium, High - Grade 3 | 0 | 1 | 0
  Sodium, High - Grade 4: number analyzed (Participants) | 133 | 130 | 132
  Sodium, High - Grade 4 | 1 | 0 | 1
  Bilirubin, High - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Bilirubin, High - Any Grade | 16 | 14 | 11
  Bilirubin, High - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Bilirubin, High - Grade 1 | 12 | 9 | 8
  Bilirubin, High - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Bilirubin, High - Grade 2 | 2 | 5 | 2
  Bilirubin, High - Grade 3: number analyzed (Participants) | 133 | 130 | 132
  Bilirubin, High - Grade 3 | 2 | 0 | 1
  Uric Acid, High - Any Grade: number analyzed (Participants) | 114 | 112 | 114
  Uric Acid, High - Any Grade | 33 | 24 | 22
  Uric Acid, High - Grade 3: number analyzed (Participants) | 114 | 112 | 114
  Uric Acid, High - Grade 3 | 33 | 24 | 22
  Total Leukocyte Count, Low - Any Grade: number analyzed (Participants) | 133 | 130 | 132
  Total Leukocyte Count, Low - Any Grade | 12 | 6 | 10
  Total Leukocyte Count, Low - Grade 1: number analyzed (Participants) | 133 | 130 | 132
  Total Leukocyte Count, Low - Grade 1 | 10 | 6 | 10
  Total Leukocyte Count, Low - Grade 2: number analyzed (Participants) | 133 | 130 | 132
  Total Leukocyte Count, Low - Grade 2 | 2 | 0 | 0

18. Secondary Outcome: Number of Participants With Vital Sign Abnormalities at Anytime Post-Baseline
Description: The number of participants with vital sign abnormalities outside of the normal upper (i.e., High) and lower limits (i.e., Low) were summarized for each parameter. The normal reference range used for each vital sign parameter was as follows: Diastolic Blood Pressure, 50-90 millimetres of mercury (mmHg); Oxygen Saturation, ≥94%; Pulse Rate, 60-100 beats per minute; Respiratory Rate, 8-20 breaths per minute; Systolic Blood Pressure, 90-140 mmHg; Temperature, 36.5-38 degrees Celsius (C). Not every vital sign abnormality qualified as an adverse event. A vital sign result was to be reported as an adverse event if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgement.
Time Frame: From Baseline up to 60 days
Population: Safety Population: participants who received at least one dose of study drug, with participants grouped according to the treatment received. Only participants with both a baseline assessment and at least one post-baseline assessment were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 133 | 130 | 132
Participants
  Diastolic Blood Pressure - Low | 23 | 23 | 21
  Diastolic Blood Pressure - High | 39 | 43 | 39
  Oxygen Saturation - Low | 112 | 107 | 105
  Pulse Rate - Low | 66 | 66 | 61
  Pulse Rate - High | 75 | 62 | 57
  Respiratory Rate - Low | 1 | 0 | 2
  Respiratory Rate - High | 108 | 104 | 103
  Systolic Blood Pressure - Low | 20 | 11 | 17
  Systolic Blood Pressure - High | 77 | 81 | 70
  Temperature - Low | 116 | 113 | 113
  Temperature - High | 13 | 10 | 14

19. Secondary Outcome: Number of Participants by the Investigator's Interpretations of Electrocardiogram Recordings at Specified Timepoints
Description: Electrocardiogram (ECG) recordings were to be performed after the participant had been resting in a supine position for at least 10 minutes if possible. The investigator's interpretation of the ECG (e.g., normal or abnormal) was recorded.
Time Frame: Baseline, Days 14 and 28, Discharge Day (up to Day 28), and Study Completion Visit (up to Day 60)
Population: Safety Population: participants who received at least one dose of study drug, with participants grouped according to the treatment received. Only participants with nonmissing assessments at a given timepoint were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
Number analyzed (Participants) | 134 | 130 | 132
Participants
  Baseline - Abnormal ECG: number analyzed (Participants) | 132 | 126 | 130
  Baseline - Abnormal ECG | 56 | 60 | 55
  Baseline - Normal ECG: number analyzed (Participants) | 132 | 126 | 130
  Baseline - Normal ECG | 76 | 66 | 75
  Day 14 - Abnormal ECG: number analyzed (Participants) | 34 | 29 | 24
  Day 14 - Abnormal ECG | 20 | 13 | 14
  Day 14 - Normal ECG: number analyzed (Participants) | 34 | 29 | 24
  Day 14 - Normal ECG | 14 | 16 | 10
  Day 28 - Abnormal ECG: number analyzed (Participants) | 15 | 5 | 7
  Day 28 - Abnormal ECG | 12 | 3 | 4
  Day 28 - Normal ECG: number analyzed (Participants) | 15 | 5 | 7
  Day 28 - Normal ECG | 3 | 2 | 3
  Discharge Day - Abnormal ECG: number analyzed (Participants) | 64 | 75 | 76
  Discharge Day - Abnormal ECG | 27 | 28 | 37
  Discharge Day - Normal ECG: number analyzed (Participants) | 64 | 75 | 76
  Discharge Day - Normal ECG | 37 | 47 | 39
  Study Completion Visit - Abnormal ECG: number analyzed (Participants) | 69 | 65 | 62
  Study Completion Visit - Abnormal ECG | 13 | 18 | 21
  Study Completion Visit - Normal ECG: number analyzed (Participants) | 69 | 65 | 62
  Study Completion Visit - Normal ECG | 56 | 46 | 40
  Study Completion Visit - Unable to Evaluate ECG: number analyzed (Participants) | 69 | 65 | 62
  Study Completion Visit - Unable to Evaluate ECG | 0 | 1 | 1

20. Secondary Outcome: Percentage of Participants Who Tested Positive for Anti-Drug Antibodies (ADAs) to MSTT1041A and UTTR1147A at Baseline and at Anytime Post-Baseline
Description: Serum samples were collected, and participants who received treatment with MSTT1041A or MSTT1041A-matched placebo were assessed for antidrug antibodies (ADAs) to MSTT1041A, while those who received UTTR1147A or UTTR1147A-matched placebo were assessed for ADAs to UTTR1147A. Participants who received placebo treatment were only assessed for the presence of ADAs at baseline. The percentage of ADA-positive participants at baseline (baseline prevalence) and after drug administration (postbaseline incidence) are summarized. When determining postbaseline incidence, participants were considered to be ADA positive if they were ADA negative or had missing data at baseline but developed an ADA response following study drug exposure (treatment-induced ADA response), or if they were ADA positive at baseline and the titer of one or more postbaseline samples was at least 0.60 titer unit greater than the titer of the baseline sample (treatment-enhanced ADA response).
Time Frame: At Baseline (pre-dose on Day 1) and post-baseline (Days 15 and 28; and discharge day and study completion [up to 60 days])
Population: The immunogenicity analysis population consisted of all participants with an evaluable baseline ADA sample and/or at least one evaluable post-baseline ADA sample. Participants who received placebo treatment were only assessed for the presence of ADAs at baseline.
Measure: Number; unit: Percentage of participants
Groups:
- MSTT1041A-Matched Placebo: Participants in this analysis group received treatment with MSTT1041A-matched placebo. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
- UTTR1147A-Matched Placebo: Participants in this analysis group received treatment with UTTR1147A-matched placebo. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
Arm/Group | MSTT1041A-Matched Placebo | MSTT1041A | UTTR1147A-Matched Placebo | UTTR1147A
Number analyzed (Participants) | 59 | 130 | 59 | 132
Percentage of participants
  ADA Positive at Baseline: number analyzed (Participants) | 59 | 117 | 59 | 126
  ADA Positive at Baseline | 3.4 | 2.6 | 1.7 | 1.6
  ADA Positive Post-Baseline (Total): number analyzed (Participants) | 0 | 104 | 0 | 107
  ADA Positive Post-Baseline (Total) |  | 2.9 |  | 0.9
  Treatment-Induced ADA Positive Post-Baseline: number analyzed (Participants) | 0 | 104 | 0 | 107
  Treatment-Induced ADA Positive Post-Baseline |  | 1.9 |  | 0.9
  Treatment-Enhanced ADA Positive Post-Baseline: number analyzed (Participants) | 0 | 104 | 0 | 107
  Treatment-Enhanced ADA Positive Post-Baseline |  | 1.0 |  | 0.0

21. Secondary Outcome: Serum Concentration of UTTR1147A at Specified Timepoints
Time Frame: For the first dose: at 0.5 hours post-dose on Day 1, on Days 2, 3, 7, and 15; and for the second dose: Days 15 (0.5 hours post-dose), 21, and 28
Population: The Pharmacokinetics (PK) analysis population for UTTR1147A consisted of participants who received at least one dose of UTTR1147A and had at least one evaluable PK concentration data point. The PK analysis population is further divided into three groups: participants who only received the first dose, participants who received both doses, and all participants who received the first dose only or both doses (from Days 1 to 15).
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Groups:
- UTTR1147A - PK Participants Who Only Received First Dose: All participants in this analysis group only received one intravenous (IV) infusion of UTTR1147A 90 micrograms/kilogram body weight (μg/kg) on Day 1. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
- UTTR1147A - PK Participants Who Received Both Doses: All participants in this analysis group received one intravenous (IV) infusion of UTTR1147A 90 micrograms/kilogram body weight (μg/kg) on Day 1 and a second IV dose of UTTR1147A 90 μg/kg on Day 15 because they remained hospitalized with a requirement for supplemental oxygen. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
- UTTR1147A - All PK Participants (First Dose Only or Both Doses), Days 1 to 15: Participants in this analysis group either received only the first dose or both doses of UTTR1147A. One intravenous (IV) infusion of UTTR1147A 90 micrograms/kilogram body weight (μg/kg) was given on Day 1, and a second IV dose of UTTR1147A 90 μg/kg was given on Day 15 if the participant remained hospitalized with a requirement for supplemental oxygen. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
Arm/Group | UTTR1147A - PK Participants Who Only Received First Dose | UTTR1147A - PK Participants Who Received Both Doses | UTTR1147A - All PK Participants (First Dose Only or Both Doses), Days 1 to 15
Number analyzed (Participants) | 105 | 25 | 130
nanograms per millilitre (ng/mL)
  Day 1, 0.5 hours post-dose: number analyzed (Participants) | 98 | 24 | 122
  Day 1, 0.5 hours post-dose | 1260 (568) | 1600 (1820) | 1320 (952)
  Day 2: number analyzed (Participants) | 96 | 23 | 119
  Day 2 | 707 (268) | 674 (372) | 700 (290)
  Day 3: number analyzed (Participants) | 84 | 24 | 108
  Day 3 | 518 (221) | 604 (222) | 537 (223)
  Day 7: number analyzed (Participants) | 46 | 24 | 70
  Day 7 | 258 (110) | 259 (109) | 258 (109)
  Day 15, pre-dose: number analyzed (Participants) | 4 | 25 | 29
  Day 15, pre-dose | 42.3 (27.8) | 88.1 (40.6) | 81.8 (41.9)
  Day 15, 0.5 hours post-dose: number analyzed (Participants) | 0 | 25 | 0
  Day 15, 0.5 hours post-dose |  | 1410 (802) |
  Day 21: number analyzed (Participants) | 1 | 14 | 0
  Day 21 | 2.69 (NA) — Standard deviation could not be calculated with data from 1 participant. | 297 (147) |
  Day 28: number analyzed (Participants) | 3 | 8 | 0
  Day 28 | 11.3 (8.89) | 173 (78.4) |

22. Secondary Outcome: Serum Concentration of MSTT1041A at Specified Timepoints
Time Frame: as for outcome 21
Population: The Pharmacokinetics (PK) analysis population for MSTT1041A consisted of participants who received at least one dose of MSTT1041A and had at least one evaluable PK concentration data point. The PK analysis population is further divided into three groups: participants who only received the first dose, participants who received both doses, and all participants who received the first dose only or both doses (from Days 1 to 15).
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Groups:
- MSTT1041A - PK Participants Who Only Received First Dose: All participants in this analysis group only received one intravenous (IV) infusion of MSTT1041A 700 milligrams (mg) on Day 1. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
- MSTT1041A - PK Participants Who Received Both Doses: All participants in this analysis group received one intravenous (IV) infusion of MSTT1041A 700 milligrams (mg) on Day 1 and a second IV dose of MSTT1041A 350 mg was given on Day 15 because they remained hospitalized with a requirement for supplemental oxygen. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
- MSTT1041A - All PK Participants (First Dose Only or Both Doses), Days 1 to 15: Participants in this analysis group either received only the first dose or both doses of MSTT1041A. One intravenous (IV) infusion of MSTT1041A 700 milligrams (mg) on Day 1, and a second IV dose of MSTT1041A 350 mg was given on Day 15 if the participant remained hospitalized with a requirement for supplemental oxygen. Study treatment was given in combination with the standard of care for COVID-19 pneumonia.
Arm/Group | MSTT1041A - PK Participants Who Only Received First Dose | MSTT1041A - PK Participants Who Received Both Doses | MSTT1041A - All PK Participants (First Dose Only or Both Doses), Days 1 to 15
Number analyzed (Participants) | 96 | 23 | 119
micrograms per millilitre (μg/mL)
  Day 1, 0.5 hours post-dose: number analyzed (Participants) | 90 | 22 | 112
  Day 1, 0.5 hours post-dose | 206 (71.1) | 227 (66.7) | 210 (70.4)
  Day 2: number analyzed (Participants) | 89 | 23 | 112
  Day 2 | 175 (49.1) | 178 (54.3) | 176 (50.0)
  Day 3: number analyzed (Participants) | 81 | 23 | 104
  Day 3 | 147 (40.1) | 135 (41.0) | 144 (40.4)
  Day 7: number analyzed (Participants) | 49 | 23 | 72
  Day 7 | 88.6 (32.3) | 83.9 (28.1) | 87.1 (30.9)
  Day 15, pre-dose: number analyzed (Participants) | 4 | 22 | 26
  Day 15, pre-dose | 32.2 (15.2) | 33.8 (17.2) | 33.5 (16.6)
  Day 15, 0.5 hours post-dose: number analyzed (Participants) | 0 | 21 | 0
  Day 15, 0.5 hours post-dose |  | 144 (48.0) |
  Day 21: number analyzed (Participants) | 0 | 9 | 0
  Day 21 |  | 45.4 (20.8) |
  Day 28: number analyzed (Participants) | 0 | 5 | 0
  Day 28 |  | 22.5 (9.17) |

ADVERSE EVENTS:
Time Frame: From Baseline until study completion/discontinuation (up to 60 days)
Arm/Group | All Placebo | MSTT1041A | UTTR1147A
All-Cause Mortality (participants affected / at risk) | 23/134 | 23/130 | 21/132
Serious Adverse Events (participants affected / at risk) | 38/134 | 38/130 | 34/132
Other Adverse Events (participants affected / at risk) | 29/134 | 42/130 | 40/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Placebo (N=134) | MSTT1041A (N=130) | UTTR1147A (N=132)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 5 (6) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 2 (2) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bacillus bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 7 (7) | 5 (5)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 3 (3) | 4 (4)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 2 (2)
Distributive shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Placebo (N=134) | MSTT1041A (N=130) | UTTR1147A (N=132)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 9 (9) | 7 (8)
Constipation (Gastrointestinal disorders) | 6 (6) | 10 (10) | 10 (10)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (8) | 9 (9) | 8 (10)
Headache (Nervous system disorders) | 4 (4) | 7 (8) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 5 (5) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4) | 9 (9)
Hypertension (Vascular disorders) | 4 (4) | 8 (8) | 2 (2)
Hypotension (Vascular disorders) | 5 (6) | 7 (8) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (3):
  • Study Protocol (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04386616/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT04386616/SAP_001.pdf
  • Informed Consent Form (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04386616/ICF_002.pdf